CLINICAL TRIAL: NCT05213507
Title: Inhaled Amikacin in Preventing Acute Exacerbation of Moderate to Very Severe Chronic Obstructive Pulmonary Disease (COPD): a Multicenter Clinical Study
Brief Title: Inhaled Amikacin in Preventing AECOPD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B2021-766; DGF501035/017 (Other: Shanghai Medical College of Fudan University)
Record Dates: First submitted 2022-01-16; First posted 2022-01-28 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: COPD; COPD Exacerbation
Keywords: Amikacin; Respiratory Tract Diseases; Anti-Bacterial Agents; Anti-Infective Agents
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Tract Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inhaled Amikacin plus Conventional Therapy (Experimental): 0.4g Amikacin sulfate injection + 5ml saline, aerosol inhalation, b.i.d., 7-10 days per month, for 3 months.
  In order to observe and cope with adverse events timely, subjects will be admitted to the ward during the course of medication.
  Subjects will take conventional therapy at the same time.
  Interventions: Drug: aerosol inhaled Amikacin Sulfate Injection; Other: conventional therapy
- Conventional Therapy (Other): According to the subjects' personal characteristics and guidance of The Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2021, the doctor in charge prescribes appropriate medication, including but not limited to bronchodilators, inhaled glucocorticoids and long-term oxygen therapy.
  Interventions: Other: conventional therapy

INTERVENTIONS:
Drug: aerosol inhaled Amikacin Sulfate Injection — 0.4g Amikacin sulfate injection + 5ml saline, aerosol inhalation, b.i.d., 7-10 days per month, for 3 months.
  Other Names: Aerosol Inhaled investigation drug
  Arms: Inhaled Amikacin plus Conventional Therapy
Other: conventional therapy — According to the personal characteristics of subjects and guidance of The Global Initiative for Chronic Obstructive Lung Disease (GOLD) 2021, the doctor in charge prescribes appropriate medication, including but not limited to bronchodilators, inhaled corticosteroids and long-term oxygen therapy.
  Other Names: Comparison Group

SUMMARY:
The underlying bacterial colonization in lower respiratory tract (LRT) of COPD patients may be related to acute exacerbation of COPD (AECOPD) and disease progression. However, there is a lack of strong evidence on the effect of LRT bacterial decolonization on COPD. This study was designed to confirm the prophylactic effect of decolonization of LRT bacteria on AECOPD and establish a novel prophylactic therapy for sable COPD.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) has become the third leading cause of death all over the world. Frequent acute exacerbations can even increase the mortality of COPD. Therefore, preventing the acute exacerbation of COPD (AECOPD) might improve prognosis.

About 74% of stable COPD patients had underlying pathogen colonization, mainly Gram-negative bacteria, in lower respiratory tract (LRT). Bacterial colonization can damage the airways of COPD patients, leading to disease progression. Further disruption of airway defense mechanisms promotes the adhesion and growth of bacteria in reverse. Eventually, a vicious circle is formed between LRT bacterial colonization and the progression of COPD. Thus, moderate to severe COPD patients were more likely to have LRT colonization, and patients with higher load of LRT bacterial colonization tended to have more frequent acute exacerbations. Decolonization of LRT bacteria may be able to control the progression of COPD and prevent AECOPD through breaking the vicious circle.

Instead of proving that long-term use of antibiotics in stable stage of COPD can prevent AECOPD, previous clinical trials have found that it can lead to the development of severe adverse reactions and the growth of LRT drug-resistant bacteria. It is probably because the main colonized LTR bacteria were not sensitive to those investigational drugs. Additionally, drugs were delivered systematically in those previous studies. Theoretically, inhalation administration can deliver the drug directly to the lungs, leading to higher drug concentrations in the lungs and less occurrence of systemic adverse reactions. Therefore, inhalation administration can well make up for the deficiencies of systematic administration. Studies on cystic fibrosis and bronchiectasis have yielded promising results of the safety and effectiveness of inhaled antibiotics for LRT bacterial decolonization. As COPD has similar manifestations to the two diseases, the promising results indicated the feasibility of decolonization of LRT bacteria to prevent AECOPD.

Previously, a multicentral clinical trial conducted by our research team preliminarily investigated whether nebulized Amikacin combined with conventional therapy could prevent AECOPD and disease progression of COPD. However, whether decolonization of LRT bacteria plays a role in these process remains unknown. The main purpose of this research is to confirm the prophylactic effect of decolonization of LRT bacteria on AECOPD and establish a novel prophylactic therapy for sable COPD.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with COPD according to GOLD 2021 (The ratio of post-bronchodilator forced expiratory volume in 1 second (FEV1) to force vital capacity (FVC) < 0.70 with the use of 400ug salbutamol)
2. Moderate to very severe airflow limitation (post-bronchodilator FEV1 < 80% of the predicted value with the use of 400ug salbutamol)
3. A documented history of at least twice AECOPD in the previous 12 months that required treatment with systemic glucocorticoids and/or antibiotics.
4. In the stable stage of COPD.
5. At least once positive result of amikacin sensitive Gram-negative bacteria by semi-quantitative sputum culture, including Pseudomonas aeruginosa, Acinetobacter baumannii, Klebsiella pneumonia, etc.
6. Written informed consent must be obtained before any assessment is performed.
7. Male or female adults aged 18-80 years.

Exclusion Criteria:

1. Patients with concomitant pulmonary disease, including bronchiectasis, interstitial lung disease, asthma, etc.
2. Patients with alpha-1 antitrypsin deficiency.
3. Patients who have had AECOPD or acute exacerbation of any other diseases that required treatment with systemic glucocorticoids and/or antibiotics in the 4 weeks prior to screening.
4. Patients with long-term oral corticosteroid use.
5. Patients with Gram-negative bacterial infection requiring systemic treatment with antibiotics against Gram-negative bacteria.
6. Patients who have participated in any interventional clinical trials in the 3 months prior to screening.
7. Patients who are allergic to amikacin or other aminoglycosides.
8. Patients who have chronic hepatic, renal and gastrointestinal abnormality or malignant tumor, except for lung cancer, which could interfere with the assessment of the efficacy and safety of the intervention.
9. Patients with mental diseases or cognitive disorders which could interfere with treatment and follow-up.
10. Patients at high risk of being lost during the 3-month treatment and the 1-year follow up.
11. Pregnant or nursing (lactating) women.
12. Patients who are in critical conditions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Time to the first COPD acute exacerbation | 15 months
  COPD acute exacerbation refers to the deterioration of daily symptoms, which requires treatment with antibiotics or systemic glucocorticoid therapy.
  The first COPD acute exacerbations was defined as the date of occurrence of the first AECOPD starting from the day of the first dose to one day after the last visit.

SECONDARY OUTCOMES:
Number of the COPD acute exacerbations | 15 months
  COPD acute exacerbation refers to the deterioration of daily symptoms, which requires treatment with antibiotics or systemic glucocorticoid therapy.
  The number of COPD acute exacerbations was defined as the number of all the AECOPD that occurs between the day of the first dose and one day after the last visit.
Load of LRT colonized potential pathogenic bacteria in induced sputum | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months
  Induced sputum represents the specimen from LRT and should be processed within 6 hours after collection. Colonized bacteria are defined by the positive results of semi-quantitative culture.
  Gram-negative bacteria, including Pseudomonas aeruginosa, Acinetobacter baumannii and Klebsiella pneumoniae, the common bacteria involved in AECOPD, are defined as potential pathogenic bacteria.
Minimum inhibitory concentration (MIC) of colonized potential pathogenic bacteria in induced sputum | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months
  Induced sputum represents the specimen from LRT and should be processed within 6 hours after collection. Colonized bacteria are defined by the positive results of semi-quantitative culture.
  Gram-negative bacteria, including Pseudomonas aeruginosa, Acinetobacter baumannii and Klebsiella pneumoniae, the common bacteria involved in AECOPD, are defined as potential pathogenic bacteria.
Microbiome in induced sputum | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months
  Induced sputum represents the specimen from LRT and should be processed within 6 hours after collection.
  Bacterial genomic DNA was isolated from sputum plugs of the same weight using the specific kits. The 16S bacterial ribosomal RNA genes were Polymerase Chain Reaction (PCR)-amplified with the appropriate controls against reagent contamination. Amplified DNA fragments were sequenced using the specific sequencing platform. Sequencing reads were processed and analyzed by the specific algorithm and software. The composition and diversity of microbiome are represented by major taxonomic groups at both phylum and genus levels. If necessary, Quantitative PCR for 16S rRNA gene will be performed to validate the results of sequencing. By using these methos, we can detect the microbiome's composition and its shift.
Forced Expiratory Volume in 1 Second | Baseline, 3 months, 15 months
  Pulmonary function assessments were performed using centralized spirometry according to international standards. FEV1 was measured 15 minutes after inhaling 400 ug salbutamol.
COPD Assessment Test (CAT) Score | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months
  The COPD Assessment Test (CAT) is an 8-item uni-dimensional measure of health status impairment in COPD, containing 6 grades from 0 to 5.
modified Medical Research Council (mMRC) scale | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months
  The modified Medical Research Council (mMRC) scale is a simple and powerful tool to evaluate the breathlessness, containing 5 grades from 0 to 4.
Number of Patients with Adverse Events, Serious Adverse Events, and Death | Baseline, 3 months, 6 months, 9 months, 12 months, 15 months
  The overall rate of adverse events reported from the day of the first dose to the last visit. Laboratory examinations, including blood routine, urine routines and hepatorenal function, and electrocardiogram are performed in each visit in order to evaluate the safety of interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Zhang, MD, PhD, Principal Investigator — Zhongshan hospital, Shanghai Medical College, Fudan University
Locations (5):
- China (5):
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Shanghai Jingan District Central Hospital, Shanghai, Shanghai Municipality
  - Shanghai Fifth People's Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Qingpu Branch of Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Wusong Branch of Shanghai Zhongshan hospital, Shanghai, Shanghai Municipality